CLINICAL TRIAL: NCT05316831
Title: Long Term Effect on Immune Response After Pneumococcal Vaccination in Patients With Chronic Lymphocytic Leukemia and Evaluation of the Effect of Revaccination
Brief Title: Immune Response After Pneumococcal Vaccination in Patient With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Principal Investigator, Bertil Uggla, Principal Investigator, Region Örebro County
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 234041
Record Dates: First submitted 2021-09-26; First posted 2022-04-07 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: CLL; Vaccine Response
MeSH Terms: interventions — 13-valent pneumococcal vaccine; 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Group A CLL patients: Previously immunized with PCV13, in this study receiving PCV13 followed by PPSV23
  Interventions: Biological: PCV13; Biological: PPSV23
- Group B (Experimental): Group B CLL patients: Previously immunized with PPSV23, in this study receiving PCV13 followed by PCV13
  Interventions: Biological: PCV13
- Group C (Active Comparator): Group C controls: Previously immunized with PCV13, in this study receiving PCV13
  Interventions: Biological: PCV13
- Group D (Active Comparator): Group C controls: Previously immunized with PPPSV23, in this study receiving PCV13
  Interventions: Biological: PCV13

INTERVENTIONS:
Biological: PCV13 — Pneumococcal polysaccharides conjugated to CRM197 carrier protein
  Other Names: Prevenar13
Biological: PPSV23 — Pneumococcal polysaccharides
  Other Names: Pneumovax23
  Arms: Group A

SUMMARY:
A randomized, multi-centre trial was conducted between 2013-2016, including 128 patients with untreated CLL from eight hematological clinics in Sweden. Vaccination with polysaccharide pneumococcal vaccine (PPSV23) or conjugated pneumococcal vaccine (PCV13) was performed and the results were published 2018. PCV13 showed a superior immune response, measured as OPA (opsonophagocytic assays) and ELISA (enzyme-linked immunosorbent assay), compared to PPSV23. Immune cells analyses after primary immunization will be performed. Between 2019-2021 a prospective follow up study was conducted of the same cohort and also included a control group. The study participants have been revaccinated with pneumococcal vaccines with the aim to evaluate the effect of repeated dose of PCV13. The antibody response (measured as titer with FMIA (fluorescent multiplexed bead-based immunoassay) and antibody function with MOPA (multiplexed opsonophagocytic assay) will be performed. Studies investigating the dynamics of immune cells before and after primary immunization and revaccination will be performed.

The study will give important answers about the optimal vaccination strategy in patients with CLL and can improve the vaccination recommendations in immunocompromised patients.

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) patients have increased risk of pneumococcal infection due to defect T-cells, complements and neutrophil/monocyte function or hypogammaglobulinaemia. Side effects of different treatment modalities add further risk of infection.

Two pneumococcal vaccines are available, non-conjugated pneumococcal polysaccharide vaccines (PPSVs) and protein-conjugated vaccines (PCVs). 23-valent Pneumovax (PPSV23) has been recommended for healthy adults to protect against invasive pneumococcal disease (IPD) in Sweden and other countries for >30 years. Patients with reduced adaptive immune function respond inadequately to PPSVs. Instead, the 13-valent Prevenar (PCV13) is recommended for a thymus-dependent immunological memory, yielding increased and persistent immune response .

In 2016, Swedish recommendations on pneumococcal vaccination of risk groups were updated, recommending PCV13 plus PPSV23 after >8 weeks, but only after individual assessment. The evidence in CLL patients is limited but the Swedish CLL-Group has adopted the recommendations. The two vaccines are administrated consecutively to broaden the protection of additional serotype. If previously PPSV23 vaccinated, the PCV13 should be given >12 months after PSV23 to avoid decreasing antibodies, i.e hyporesponse, but this is not studied in CLL patients.

Between 2013-2016, the investigators conducted a phase III trial at 8 hematological clinics in Sweden, including 126 untreated CLL patients, randomized to PCV13 (n=63) or PPSV23 (n=63) . The immune response was analyzed in terms of antibody induction and functionality, measured by enzyme-linked immunosorbent assay (ELISA) and opsonophagocytosis assay (OPA), respectively. The proportion of responding patients was larger for PCV13 than for PPSV23 after 4 weeks (40% vs. 22%, p=0.03) and 6 months (33% vs. 17%, p=0.04).

This study aims to investigate the persistent antibody protection in CLL patients 4-6 years after vaccination with PCV13 (n=63) vs PPSV23 (n=63), and the effect of revaccination with PCV13 in both groups. Also, the aim is to study if a repeated dose of PCV13 results in improved response, similar to controls after one dose of PCV13, and compared to PCV13 plus PPSV23 revaccination. Secondly, the study investigates the effect of pneumococcal vaccination on incidence of pneumococcal infection and colonization. A control group (N=32) has been included. Peripheral blood mononuclear cell (PBMC) have been collected and further studies on the dynamics of immune cells and cytokines before and after primary immunization and revaccination with polysaccharide vaccines and conjugated vaccines will be investigated.

A sub study was initiated february 2021 in the same cohort for sampling after vaccination against SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2) in the same study cohort, enabling comparison of immune response after administrating mRNA (messenger ribonucleic acid) vaccines.

ELIGIBILITY:
Inclusion Criteria:

CLL patients earlier included in the Pneumococcal vaccination study 0887x1-20003 (EudraCT No: 2009-012642-22), who have received either PCV13 or PPSV23 are eligible for evaluation

Exclusion Criteria:

1. Patients receiving high dose corticosteroids ( ≥20 mg Prednisolone) or other immunosuppressive drugs that is not part of active CLL treatment (criteria for inclusion after discontinuing high dose corticosteroid treatment, see section 7.3)
2. Patients who have had an allergic reaction to any vaccination in the past
3. Patients with a positive DAT (Direct Antiglobulin Test) or known present or previous hemolysis, ITP (immune thrombocytopenia) and Guillain-Barre
4. Patients failing to give informed consent
5. Patients with ongoing immunoglobulin therapy
6. Patients with known HIV infection
7. Patients who have received a pneumococcal vaccine outside the study protocol within the last 12 months
8. Active febrile infection
9. Increased bleeding risk due to severe thrombocytopenia or other coagulopathies that would, in the opinion of the investigator, contraindicate intramuscular injection (for treatment with oral anticoagulation therapy, see section 7.3) -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Immune response 3-5 years after primary vaccination with a single dose of 13-valent pneumococcal conjugated vaccine (PCV13, Prevenar13®) or conventional 23-valent capsular polysaccharide vaccine (PPSV23, Pneumovax®) | 3-5 years after vaccination
  The long-term immune response, comparing the two vaccines PCV13 and PPSV23, 3-5 years after vaccination, measured as the proportion of subjects with a positive vaccination response in each of the two groups. A positive vaccination response is defined as a post vaccination OPA titer ≥ (LLOQ) in 8 of the 12 serotypes common for PCV13 and PPSV23 in serum collected
Change in immune response after revaccination. | Before and 8, 16 and 52 weeks after first revaccination
  The change in immune response 8,16 and 52 weeks after first revaccination with PCV 13 (followed by a second revaccination, 8 weeks after first revaccination, with either PPSV23 (group A) or PCV13 (group B). Immune response is measured as the proportion of subjects with a positive vaccination response pre- and post- revaccination.

SECONDARY OUTCOMES:
Prevalence of pneumococcal colonization | Before and 8, 16 and 52 weeks after first revaccination
  To study the incidence of pneumococcal colonization by naso-pharyngeal culturing nasopharyngeal swabs at inclusion after 8 weeks, 16 weeks and 12 months.
Effect of pneumococcal revaccination on T- and B-cell subsets | Before, 7 days and 8 weeks after every revaccination. Twelve months after first revaccination
  Dynamics of T- and B-cell subsets before and after revaccination will be explored using flow cytometry to determine the proportions of different B- and T-cell subsets
Antibody response after vaccination with PPSV23, PCV13 and mRNA vaccine | Before, 4-8 weeks after every vaccination and 12 months after first pneumococcal revaccination and second mRNA vaccination
  Antibody titers measured with FMIA regarding pneumococcal antibodies and Diasorins SARS-CoV-2 TrimericS IgG test (COV2TG) regarding Covid-19 antibodies, comparing antibody response to polysaccharide vaccine, conjugated vaccine and mRNA vaccine
Incidence of invasive pneumococcal disease (IPD) | From the initial vaccination to maximum five years after the first dose of revaccination
  To determine the incidence of IPD among the study participants by collecting data from medical records
Effect of pneumococcal revaccination on cytokine levels | Before and 8, 16 and 52 weeks after first revaccination
  Investigate the dynamics of cytokine levels before and after revaccination determined by multiplex immunoassays
Immune cell response after vaccination with PPSV23, PCV13 and mRNA vaccine | Before, 4-8 weeks afte0r every vaccination and 12 month after first pneumococcal revaccination and second mRNA vaccination
  Dynamic of T- and B-cell subsets before and after vaccination with polysaccharide vaccine, conjugated vaccine and mRNA vaccine using flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Bertil Uggla, Md, PhD, Principal Investigator — Universitetssjukhuset Örebro
Locations (1):
- Magdalena Kättström, Örebro, Sweden

REFERENCES:
- [Derived] Kattstrom M, Uggla B, Virta C, Melin M, Ekstrom N, Magnuson A, Andersson PO, Hammarlund Y, Lockmer S, Nilsson I, Roth D, Svensson M, Tolf T, Kimby E, Noren T, Athlin S. Revaccination with pneumococcal conjugate vaccine five years after primary immunization improves immunity in patients with chronic lymphocytic leukemia. Haematologica. 2025 Aug 1;110(8):1774-1785. doi: 10.3324/haematol.2024.286942. Epub 2025 Mar 6. PMID 40045895